CLINICAL TRIAL: NCT00694850
Title: A Multi-center, Non-randomized, Non Blinded, Non-controlled Study to Investigate the Impact of Multiple Doses of BAY63-2521 on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Patients With Interstitial Lung Disease Associated Pulmonary Hypertension.
Brief Title: Impact of Multiple Doses of BAY63-2521 on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Patients With Interstitial Lung Disease (ILD) Associated Pulmonary Hypertension (PH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12916; 2023-507526-17-00 (Other: CTIS (EU)); 2007-003928-37 (EudraCT Number)
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypertension, Pulmonary
Keywords: Interstitial lung disease associated pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY63-2521).

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521). — BAY63-2521 will be up-titrated from 1,0 mg TID to 2,5 mg TID

SUMMARY:
The purpose of this study is to assess multiple ascending doses of a new drug (BAY63-2521) given orally, to evaluate if it is safe and can help to improve the well-being, symptoms (e.g. disturbed breathing) and outcome of pulmonary hypertension associated with lung fibrosis. Patients living with pulmonary hypertension associated with interstitial lung disease have a risk of increased number of hospitalisations because of worsening of their condition. Until now there is no approved medication for this disease. The current treatment of pulmonary hypertension associated with interstitial lung disease consists: of oxygen and medical treatment with vasodilators, e.g. so-called Calcium-antagonists. Therefore, there is a need for new drugs in the treatment of pulmonary hypertension associated with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an interstitial lung disease (usual interstitial pneumonia [UIP], nonspecific interstitial pneumonia [NSIP] or sarcoidosis) with high resolution CT and a total lung capacity (TLC) ≤ 90% or scleroderma associated pulmonary arterial hypertension (PAH) with total lung capacity (TLC) ≤ 80%.
* Interstitial lung disease (ILD) must have been stable for at least 3 months (decrease in forced vital capacity (FVC)< 10% and diffusing capacity of lung for carbon monoxide (DLco) < 15 % in 3 months), i.e. no significant changes in pulmonary function testing and stable medication in terms of ILD (e.g., corticosteroids, immunosuppressants)
* Mean pulmonary vascular resistance (PVR) > 400 dyne sec cm-5 or mean pulmonary arterial pressure (PAP mean) > 30 mmHg
* Pulmonary capillary wedge pressure (PCWP) < 15 mmHg
* Hemodynamic parameters at baseline (PAP, PCWP, cardiac output [CO], systemic mean arterial pressure [SAP])
* High resolution computer tomography (HRCT) (should not be older than 12 months prior start of the study)
* Heart rate > 55 beats per minute (BPM) and < 105 BPM at rest
* Systolic blood pressure (SBP) > 90 mmHg
* World Health Organisation (WHO) functional class II, III and IV
* 6 Minute Walking Test (6MWT) > 100m and < 450 m
* Stable controlled arterial hypertension according to current guidelines
* Women of childbearing potential will be included in the study if the pregnancy test is negative and combination of condoms with a safe and highly effective contraception method (hormonal contraception with implants or combined oral contraceptives, certain intra-uterine devices [IUDs]) is granted.

Exclusion Criteria:

* Co-medication:

  * Patients pretreated with specific medication for pulmonary arterial hypertension (PAH) like endothelin receptor antagonists, prostaglandins or phosphodiesterase type 5 (PDE 5) blockers are excluded from the trial.
  * Requirement for concomitant use of nitrates are contraindicated.
* Pre-existing clinically relevant lung disease other than ILD including.

  * Bronchial asthma and Chronic Obstructive Pulmonary Disease (COPD) with a forced expiratory volume in one second (FEV1)/FVC <60% pred., active tuberculosis
  * Pulmonary hypertension of another WHO group (I, II, IV and V)
  * Severe congenital abnormalities of the lungs, thorax and diaphragm
  * Clinical or radiological evidence of a pulmovenoocclusive disease (PVOD)
* Systemic hemodynamics

  * Acute or severe chronic left heart failure (ejection fraction (EF) < 50%)
  * Severe coronary artery disease (CAD; EF < 50%); CAD patients must be asymptomatic and stable
  * Congenital or acquired valvular or myocardial disease if clinically significant apart from tricuspid valvular insufficiency due to pulmonary hypertension
* Pulmonary function

  * TLC predicted < 30%
  * FEV1 (related to FVC) < 60% predicted
* Blood gases at room air

  * Arterial partial carbon dioxide pressure (Pa CO2) > 45 mmHg
  * Arterial partial oxygen pressure (Pa O2) < 50 mmHg at O2 supply >/= 4 L/min
* Peripheral organ function

  * Moderate or severe hepatic insufficiency (Child-Pugh Class Band C and/or total bilirubin > 2.5 mg/dl (0.043 mmol/L); and/or hepatic transaminases >3 upper limit normal [ULN])
  * Moderate or severe renal insufficiency (creatinine > 2 mg/dl) or creatinine clearance according to Cockroft-Gault formula < 35 mL/ min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08-02 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 12 weeks treatment

SECONDARY OUTCOMES:
Pharmacokinetics | at every study visit except at run-in and Follow-up
  The assessment will be stopped after protocol amendment 4, which was effective since Jan 06, 2014
6-Minute Walk Test | at every study visit except at Follow-up
Modified borg scale | at every study visit except at Follow-up
  The assessment will be stopped after protocol amendment 4, which was effective since Jan 06, 2014
Quality of life assessments | at baseline, after 6 weeks, after 12 weeks, Follow-up and at each visit during long term extension phase
  The assessment will be stopped after protocol amendment 4, which was effective since Jan 06, 2014
Hemodynamic parameters | optional after 12weeks
Laboratory Parameters | at each study visit during run-in and treatment phase and long term extension
  The assessment will be stopped after protocol amendment 4, which was effective since Jan 06, 2014
Electrocardiogram (ECG) | at each study visit during run-in and treatment phase and long term extension
  The assessment will be stopped after protocol amendment 4, which was effective since Jan 06, 2014
Blood pressure and heart rate | at each study visit during run-in and treatment phase and long term extension

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Germany (5):
  - München, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Homburg, Saarland
  - Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Result] Hoeper MM, Halank M, Wilkens H, Gunther A, Weimann G, Gebert I, Leuchte HH, Behr J. Riociguat for interstitial lung disease and pulmonary hypertension: a pilot trial. Eur Respir J. 2013 Apr;41(4):853-60. doi: 10.1183/09031936.00213911. Epub 2012 Aug 30. PMID 22936711
- See also: Click here and search for drug information provided by the FDA. — https://www.fda.gov/drugs/drug-safety-and-availability/drug-safety-communications
- See also: Click here and search for information on any recalls, market or product safety alerts by the FDA which might have occurred with this product. — https://www.fda.gov/safety/medwatch-fda-safety-information-and-adverse-event-reporting-program